CLINICAL TRIAL: NCT07149064
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Efficacy and Safety of Chronic Exposure to Nextida GC-B on Glycemic Control in Adults With Normoglycemia or Prediabetes
Brief Title: Effect of Chronic Exposure to Nextida GC-B on Glycemic Control in Adults With Normoglycemia or Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25RSCFA01
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Normoglycemia; Prediabetes; Glycemic Control
Keywords: Nextida GC-B; glycemic control; normoglycemia; Prediabetes; postprandial glycemic control
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nextida GC-B (Experimental): This group receives one liquid shot of 5 g Nextida GC-B approximately 30 minutes before their two main meals (breakfast and lunch or breakfast and dinner) daily.
  Interventions: Dietary Supplement: Nextida GC-B
- Placebo (Placebo Comparator): This group receives one liquid shot of placebo approximately 30 minutes before their two main meals (breakfast and lunch or breakfast and dinner) daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nextida GC-B — One liquid shot contains 5 g of collagen hydrolysate.
  Arms: Nextida GC-B
Other: Placebo — One liquid shot contains non-active ingredients in Nextida GC-B (water, Erythritol, Citric Acid, DL-Malic Acid, Natural Apples Flavor, Steviol Glycosides).
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of Nextida GC-B on glycemic control in adults with normoglycemia and prediabetes. The main question it aims to answer is:

What is the difference in change in postprandial glycemic control from baseline at Day 90 between Nextida GC-B and placebo as assessed by glucose incremental AUC (iAUC 0-180 min).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years and older
2. BMI of 25 to 34.9 kg/m2, inclusive
3. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   2. Double-barrier method
   3. Intrauterine devices
   4. Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   5. Vasectomy of partner at least 6 months prior to screening
   6. Abstinence and agrees to use contraception if planning on becoming sexually active during the study
4. Individuals with normoglycemia (HbA1c ≤5.9%) or prediabetes (HbA1c 6.0 to ≤6.4%) at screening
5. Stable body weight defined as a <5% change in body weight in the three months prior to baseline as assessed by the Qualified Investigator (QI)
6. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, sleep, and skin, nail and hair habits) as much as possible throughout the study
7. Willingness to complete questionnaires, records and diaries associated with the study, comply with continuous glucose monitor (CGM) device instructions, and complete all clinic visits
8. Provided voluntary, written, informed consent to participate in the study
9. Healthy as determined by medical history and laboratory results as assessed by QI

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational product, placebo or standardized meal ingredients
3. Metal implants or other physical characteristics/limitations that may affect DEXA scan results as assessed by the QI
4. Poor venous access as assessed by the QI
5. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Section 7.3)
6. Unstable metabolic disease or chronic diseases as assessed by the QI
7. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
8. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
9. Type I or Type II diabetes
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
16. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
17. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
18. Use of medical cannabinoid products
19. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
20. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
21. Alcohol intake average of >2 standard drinks per day as assessed by the QI
22. Alcohol or drug abuse within the last 12 months
23. Clinically significant abnormal laboratory results at screening as assessed by the QI
24. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
25. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
26. Individuals who are unable to give informed consent
27. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The difference in change in postprandial glycemic control between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in postprandial glycemic control from baseline at Day 90 between Nextida GC-B and placebo as assessed by glucose incremental area under the curve (AUC) (iAUC 0-180 min).
The difference in change in glycated hemoglobin (HbA1c) and glucose variability from baseline at Day 90 between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in glycated hemoglobin (HbA1c) and glucose variability between Nextida GC-B and placebo

SECONDARY OUTCOMES:
The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax) | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax)
The difference in change between Nextida GC-B and placebo in postprandial glucose maximum concentration (Cmax) | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial glucose maximum concentration (Cmax)
The difference in change between Nextida GC-B and placebo in postprandial insulin iAUC | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial insulin iAUC
The difference in change between Nextida GC-B and placebo in postprandial insulin Tmax | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial insulin Tmax
The difference in change between Nextida GC-B and placebo in postprandial insulin Cmax | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial insulin Cmax
The difference in change between Nextida GC-B and placebo in postprandial redox status as assessed by reduced and oxidized glutathione ratio (GSH/GSSG) | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in redox status as assessed by reduced and oxidized glutathione ratio (GSH/GSSG)
The difference in change between Nextida GC-B and placebo in postprandial redox status as assessed by reduced and oxidized glutathione ratio (GSH/GSSG) | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in post prandial redox status as assessed by reduced and oxidized glutathione ratio (GSH/GSSG)
The difference in change between Nextida GC-B and placebo in postprandial gut hormones as assessed by glucagon-like peptide-1 (GLP-1) and gastric inhibitory polypeptide (GIP) | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in post prandial gut hormones as assessed by glucagon-like peptide-1 (GLP-1) and gastric inhibitory polypeptide (GIP)
The difference in change between Nextida GC-B and placebo in postprandial hunger. | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial hunger as assessed by hunger and satiety visual analogue scales (VAS). One a scale of 1 to 7, with 1 being "not hungry at all" and 7 being "very very hungry"
The difference in change between Nextida GC-B and placebo in postprandial satiety. | Day 0 to 90
  The difference in change from baseline at Day 90 between Nextida GC-B and placebo in postprandial satiety as assessed by hunger and satiety visual analogue scales (VAS). One a scale of 1 to 7, with 1 being "not at all satisfactory and 7 being "completely satisfactory".
The difference in change from baseline between Nextida GC-B and placebo in fasting blood glucose | Day 0 to 1
  The difference in change between Nextida GC-B and placebo in fasting blood glucose
The difference in change from baseline between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG | Day 0 to 1
  The difference in change between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG
The difference in change from baseline between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP | Day 0 to 1
  The difference in change between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP
The difference in change from baseline between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. | Day 0 to 1
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. On a scale of 1 indicating "not hungry at all" to 10 indicating "extremely hungry".
The difference in change from baseline between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. | Day 0 to 1
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. On a scale of 1 indicating "not satisfied at all" to 10 indicating "extremely satisfied".
The difference in change in markers of protein glycation between Nextida GC-B and placebo in glycated hemoglobin (HbA1c) | Day 0 to 30
  The difference in change in markers of protein glycation from baseline at Day 30 between Nextida GC-B and placebo in glycated hemoglobin (HbA1c)
The difference in change in markers of protein glycation between Nextida GC-B and placebo in glycated albumin (GA) | Day 0 to 30
  The difference in change in markers of protein glycation from baseline at Day 30 between Nextida GC-B and placebo in glycated albumin (GA)
The difference in change in markers of protein glycation between Nextida GC-B and placebo in glycated albumin (GA) | Day 0 to 90
  The difference in change in markers of protein glycation from baseline at Day 90 between Nextida GC-B and placebo in glycated albumin (GA)
The difference in change in lipid profile between Nextida GC-B and placebo. | Day 0 to 30
  The difference in change in lipid profile between Nextida GC-B and placebo from baseline at Day 30.
The difference in change in lipid profile between Nextida GC-B and placebo. | Day 0 to 90
  The difference in change in lipid profile between Nextida GC-B and placebo from baseline at Day 90.
The difference in change in body weight between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in body weight from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in body weight between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body weight from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in body mass index (BMI) between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in body mass index (BMI) from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in body mass index (BMI) between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body mass index (BMI) from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in body composition between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body composition (fat mass (kg and % of total weight) from baseline at Day 90 between Nextida GC-B and placebo as assessed by DEXA scan.
The difference in change in Interleukin-6 (IL-6) between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in Interleukin-6 (IL-6) from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in Interleukin-6 (IL-6) between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in Interleukin-6 (IL-6) from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in C-reactive protein (CRP) between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in C-reactive protein (CRP) from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in C-reactive protein (CRP) between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in C-reactive protein (CRP) from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in Tumor necrosis factor-α (TNF-α) between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in Tumor necrosis factor-α (TNF-α) from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in Tumor necrosis factor-α (TNF-α) between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in Tumor necrosis factor-α (TNF-α) from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in interferon-gamma (IFN-ɣ) between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in interferon-gamma (IFN-ɣ) from baseline at Day 30 between Nextida GC-B and placebo.
The difference in change in interferon-gamma (IFN-ɣ) between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in interferon-gamma (IFN-ɣ) from baseline at Day 90 between Nextida GC-B and placebo.
The difference in change in quality of life between Nextida GC-B and placebo | Day 0 to 30
  The difference in change in quality of life from baseline at Day 30 between Nextida GC-B and placebo as assessed by the RAND SF-36 Questionnaire. On a scale of 1 to 5, with higher scores meaning a worse outcome.
The difference in change in quality of life between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in quality of life from baseline at Day 90 between Nextida GC-B and placebo as assessed by the RAND SF-36 Questionnaire. On a scale of 1 to 5, with higher scores meaning a worse outcome.
The difference in change in product perception between Nextida GC-B and placebo | Day 0 to 90
  The difference in product perception at Day 90 between Nextida GC-B and placebo as assessed by the Product Perception Questionnaire (PPQ). Product perception is not scored on a scale.
The difference in change in measures of skin health between Nextida GC-B and placebo including elasticity | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including elasticity as assessed by Corneometer®
The difference in change in measures of skin health between Nextida GC-B and placebo including elasticity | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including elasticity as assessed by Cutometer®
The difference in change in measures of skin health between Nextida GC-B and placebo including wrinkles, texture, and age spots as assessed by Visia® | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including wrinkles, texture, and age spots as assessed by Visia®
The difference in change in measures of skin health between Nextida GC-B and placebo including subjective skin quality as assessed by Modified Skin Self-Assessment Questionnaire. | Day 0 to 30
  The difference in change in measures of skin health from baseline at Day 30 between Nextida GC-B and placebo including subjective skin quality as assessed by Modified Skin Self-Assessment Questionnaire. No numbering scale is used for this assessment. Scale is from "very satisfied" to "very Unsatisfied".
The difference in change in measures of skin health between Nextida GC-B and placebo including subjective skin quality as assessed by Modified Skin Self-Assessment Questionnaire. | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including subjective skin quality as assessed by Modified Skin Self-Assessment Questionnaire.
The difference in change in nail health between Nextida GC-B and placebo as assessed by the Modified Nail Self-Assessment Questionnaire | Day 0 to 30
  The difference in change in nail health from baseline at Day 30 between Nextida GC-B and placebo as assessed by the Modified Nail Self-Assessment Questionnaire. No numbering scale is used for this assessment. Scale is from "very satisfied" to "very Unsatisfied".
The difference in change in nail health between Nextida GC-B and placebo as assessed by the Modified Nail Self-Assessment Questionnaire | Day 0 to 90
  The difference in change in nail health from baseline at Day 90 between Nextida GC-B and placebo as assessed by the Modified Nail Self-Assessment Questionnaire. No numbering scale is used for this assessment. Scale is from "very satisfied" to "very Unsatisfied".
The difference in change in hair health between Nextida GC-B and placebo as assessed by the Modified Hair Self-Assessment Questionnaire | Day 0 to 30
  The difference in change in hair health from baseline at Day 30 between Nextida GC-B and placebo as assessed by the Modified Hair Self-Assessment Questionnaire. No numbering scale is used for this assessment. Scale is from "very satisfied" to "very Unsatisfied".
The difference in change in hair health between Nextida GC-B and placebo as assessed by the Modified Hair Self-Assessment Questionnaire | Day 0 to 90
  The difference in change in hair health from baseline at Day 90 between Nextida GC-B and placebo as assessed by the Modified Hair Self-Assessment Questionnaire. No numbering scale is used for this assessment. Scale is from "very satisfied" to "very Unsatisfied".
The difference in change in body composition between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body composition (lean mass (kg and % of total weight)) from baseline at Day 90 between Nextida GC-B and placebo as assessed by DEXA scan.
The difference in change in body composition between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body composition (android fat (%)) from baseline at Day 90 between Nextida GC-B and placebo as assessed by DEXA scan.
The difference in change in body composition between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in body composition gynoid fat (%) from baseline at Day 90 between Nextida GC-B and placebo as assessed by DEXA scan.
The difference in change in body composition between Nextida GC-B and placebo | Day 0 to 90
  The difference in change in android/gynoid fat ratio from baseline at Day 90 between Nextida GC-B and placebo as assessed by DEXA scan.
The difference in change in measures of skin health between Nextida GC-B and placebo including hydration | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including hydration as assessed by Corneometer®
The difference in change in measures of skin health between Nextida GC-B and placebo including firmness | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including firmness as assessed by Corneometer®
The difference in change in measures of skin health between Nextida GC-B and placebo including firmness | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including firmness as assessed by Cutometer®
The difference in change in measures of skin health between Nextida GC-B and placebo including hydration | Day 0 to 90
  The difference in change in measures of skin health from baseline at Day 90 between Nextida GC-B and placebo including hydration as assessed by Cutometer®
The difference in change in postprandial glycemic control | Day 0 to 1
  The difference in change in postprandial glycemic control between Nextida GC-B and placebo in glucose incremental AUC (iAUC 0-180 min)
The difference in change in postprandial glycemic control | Day 0 to 30
  The difference in change in postprandial glycemic control between Nextida GC-B and placebo in glucose incremental AUC (iAUC 0-180 min)
The difference in change in postprandial glycemic control | Day 1 to 30
  The difference in change in postprandial glycemic control between Nextida GC-B and placebo in glucose incremental AUC (iAUC 0-180 min)
The difference in change in postprandial glycemic control | Day 1 to 90
  The difference in change in postprandial glycemic control between Nextida GC-B and placebo in glucose incremental AUC (iAUC 0-180 min)
The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax) | Day 0 to 1
  The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax)
The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax) | Day 0 to 30
  The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax)
The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax) | Day 1 to 30
  The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax)
The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax) | Day 1 to 90
  The difference in change between Nextida GC-B and placebo in postprandial glucose time to maximum concentration (Tmax)
The difference in change in glucose variability between Nextida GC-B and placebo as assessed by a continuous glucose monitor (CGM) | Day 0 to 7
  The difference in change in glucose variability between Nextida GC-B and placebo as assessed by a continuous glucose monitor (CGM)
The difference in change from baseline between Nextida GC-B and placebo in fasting blood glucose | Day 0 to 30
  The difference in change between Nextida GC-B and placebo in fasting blood glucose
The difference in change from baseline between Nextida GC-B and placebo in fasting blood glucose | Day 0 to 90
  The difference in change between Nextida GC-B and placebo in fasting blood glucose
The difference in change between Nextida GC-B and placebo in fasting insulin | Day 0 to 1
  The difference in change between Nextida GC-B and placebo in fasting insulin
The difference in change between Nextida GC-B and placebo in fasting insulin | Day 0 to 30
  The difference in change between Nextida GC-B and placebo in fasting insulin
The difference in change between Nextida GC-B and placebo in fasting insulin | Day 0 to 90
  The difference in change between Nextida GC-B and placebo in fasting insulin
The difference in change from baseline between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG | Day 0 to 30
  The difference in change between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG
The difference in change from baseline between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG | Day 0 to 90
  The difference in change between Nextida GC-B and placebo in fasting Redox status as assessed by GSH/GSSG
The difference in change from baseline between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP | Day 0 to 30
  The difference in change between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP
The difference in change from baseline between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP | Day 0 to 90
  The difference in change between Nextida GC-B and placebo in fasting gut hormones as assessed by GLP-1 and GIP
The difference in change from baseline between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. | Day 0 to 30
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. On a scale of 1 indicating "not hungry at all" to 10 indicating "extremely hungry".
The difference in change from baseline between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. | Day 0 to 90
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting hunger as assessed by hunger and satiety VAS. On a scale of 1 indicating "not hungry at all" to 10 indicating "extremely hungry".
The difference in change from baseline between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. | Day 0 to 30
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. On a scale of 1 indicating "not satisfied at all" to 10 indicating "extremely satisfied".
The difference in change from baseline between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. | Day 0 to 90
  The difference in change from baseline at Days 30 and 90 between Nextida GC-B and placebo in fasting satiety as assessed by hunger and satiety VAS. On a scale of 1 indicating "not satisfied at all" to 10 indicating "extremely satisfied".

OTHER OUTCOMES:
Clinically relevant changes in blood pressure (BP) after supplementation. | Day 0 to 90
  Clinically relevant changes in blood pressure (BP) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event.
Clinically relevant changes in heart rate after supplementation. | Day 0 to 90
  Clinically relevant changes in heart rate after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event.
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (aspartate aminotransferase (AST)). Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (alanine aminotransferase (ALT)) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (total bilirubin) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (creatinine) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (electrolytes (Na, K, Cl) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in clinical chemistry | Day 0 to 90
  Clinically relevant changes in clinical chemistry (estimated glomerular filtration rate (eGFR)) after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event
Clinically relevant changes in complete blood count after supplementation | Day 0 to 90
  Clinically relevant changes in complete blood count after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada